CLINICAL TRIAL: NCT00776347
Title: Donepezil Therapy and Changes of Symptoms and Glucose Metabolism in Patients With Dementia With Lewy Bodies (DLB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Responsible Party: Principal Investigator, Hiroaki Kazui, M.D,Ph.D, Osaka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSK-08096
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Dementia With Lewy Bodies (DLB)
Keywords: Dementia with Lewy bodies (DLB); FDG-PET
MeSH Terms: conditions — Lewy Body Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- donepezil (Experimental)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Dosage: 3mg PO/day for the first 2 weeks and 5mg PO/day for the next 14 weeks Duration: 16 weeks
Drug: Donepezil

SUMMARY:
The purpose of this study is to evaluate change of cerebral glucose metabolism by donepezil therapy and to associate change of glucose metabolism and symptoms.

ELIGIBILITY:
Inclusion Criteria:

DLB patients:

* who fulfill the diagnostic criteria of DLB
* 60 to 85 years old
* right-handed
* Clinical Dementia Rating (CDR) ≧ 0.5
* Mini Mental State Examination (MMSE) score from 10 to 26

Normal Controls:

* who are independent
* who have no subjective or objective cognitive impairment
* 60 to 85 years old
* right-handed
* MMSE score over 24

Exclusion Criteria:

DLB patients:

* who have diabetes mellitus
* who have pathological change on MRI other than brain atrophy
* who have complication or history of dementia other than DLB, psychiatric disease, and physical disorder that affect brain function
* who have severe complication of cardiovascular, hepatic, renal, or other diseases unable to secure the safety
* who have severe digestive ulcus
* who have severe bronchitic asthma or obstructive lung disease
* who have no caregiver who knows patient's condition well

Normal Controls:

* who have diabetes mellitus
* who have taken donepezil before
* who have abnormal findings on MRI
* who have complication or history of brain injury, psychiatric disease, and physical disorder that affect brain function

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
FDG-PET | 14 weeks

SECONDARY OUTCOMES:
Cognitive function, psychiatric symptoms, global clinical function, and burden of caregiver | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Kazui, MD, PhD, Principal Investigator — Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

REFERENCES:
- [Derived] Kanemoto H, Kazui H, Adachi H, Yoshiyama K, Wada T, Nomura KT, Shimosegawa E, Ikeda M. Thalamic pulvinar metabolism, sleep disturbances, and hallucinations in dementia with Lewy bodies: Positron emission tomography and actigraphy study. Int J Geriatr Psychiatry. 2020 Aug;35(8):934-943. doi: 10.1002/gps.5315. Epub 2020 Jun 8. PMID 32346907
- See also: Related Info — http://www.med.osaka-u.ac.jp/index-e.html